CLINICAL TRIAL: NCT07278843
Title: Natural History of Photoreceptor Degeneration Related to USH1B: Clinical Parameters and Validation of Functional Vision Tests in MYO7A
Brief Title: Natural History of Photoreceptor Degeneration in USH1B: Clinical Parameters and Validation of Functional Vision Tests in MYO7A
Acronym: MYO7A
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Other Study IDs: P25-01
Record Dates: First submitted 2025-07-23; First posted 2025-12-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Usher Syndrome
Keywords: Retina; Genetic mutation; Inherited disease; Retinis pigmentosa; Usher syndrome
MeSH Terms: conditions — Usher Syndromes; Genetic Diseases, Inborn | interventions — Vision Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pediatric Cohort 1: 3-5 years old
  Interventions: Diagnostic Test: Vision tests; Diagnostic Test: Retinal imaging
- Pediatric Cohort 2: 6-13 years old
  Interventions: Diagnostic Test: Vision tests; Diagnostic Test: Retinal imaging
- Adult Cohort: 14-75 years old
  Interventions: Diagnostic Test: Vision tests; Diagnostic Test: Retinal imaging; Diagnostic Test: Questionnaires; Diagnostic Test: Streetlab performance tests

INTERVENTIONS:
Diagnostic Test: Vision tests — Standardized assessments of visual function including best corrected visual acuity (BCVA), low vision acuity (BRVT), low luminance visual acuity (LLVA), color and contrast sensitivity tests, visual field measurements, and electroretinography (ERG) to evaluate retinal function.
Diagnostic Test: Retinal imaging — Advanced imaging techniques such as optical coherence tomography (OCT), fundus autofluorescence (FAF), and OCT angiography (OCT-A) are used to visualize retinal structure and detect abnormalities.
Diagnostic Test: Questionnaires — Patient-reported outcome measures including the Michigan Vision-Related Anxiety Questionnaire (MAVQ) and the Michigan Retinal Degeneration Questionnaire (MRDQ) assess the psychological and quality-of-life impacts of retinal degeneration.
  Groups: Adult Cohort
Diagnostic Test: Streetlab performance tests — Virtual reality-based functional tests evaluating mobility (MOST-VR) and visual search performance (VR-ViSA) to assess real-world vision-related abilities.
  Groups: Adult Cohort

SUMMARY:
Inherited retinal diseases (IRDs) are a group of degenerative disorders that cause progressive vision loss. Retinitis pigmentosa (RP) is the most common form, with a global prevalence of approximately 1 in 4,500. About 20-30% of these cases are syndromic, most notably Usher syndrome (USH), which combines hearing loss with visual impairment. Usher syndrome type 1 (USH1), the most severe form, presents at birth with profound sensorineural hearing loss, vestibular areflexia, and early-onset retinal degeneration. Biallelic mutations in the MYO7A gene, which define the USH1B subtype, account for 70% of USH1 cases. There is currently no treatment available for this serious condition. The objective of the study is to characterize the natural history of retinal degeneration in USH1B patients and to validate functional vision tests using virtual reality and patient-reported outcome questionnaires.

DETAILED DESCRIPTION:
Inherited retinal diseases (IRDs) are a heterogeneous group of disorders that gradually lead to severe visual impairment, with limited therapeutic options available. Rod dystrophy, also known as retinitis pigmentosa (RP), is the most common form of IRD, with an estimated global prevalence of 1 in 4,500. Approximately 20% to 30% of rod-cone dystrophy cases are syndromic, with Usher syndrome (USH) being the most frequent. USH has an estimated prevalence of 1 to 4 per 25,000 individuals and accounts for 50% of all cases of deafblindness and 3% to 6% of all cases of childhood deafness.

Usher syndrome type 1 (USH1) is the most severe form of the disease. It typically presents with congenital severe-to-profound sensorineural hearing loss, vestibular areflexia, and early-onset rod-cone dystrophy, usually within the first decade of life. Mutations in nine different genes have been associated with USH1, among which biallelic mutations in the MYO7A gene account for approximately 70% of cases. This specific subtype is referred to as USH1B.

There is currently no approved treatment for USH1B, representing a significant unmet medical need for this severe condition.

Objectives:

1. To study the natural history of retinal degeneration in a large USH1B patient cohort.
2. To validate functional vision tests based on virtual reality, along with two patient-reported outcome questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 3 years old;
* Have a clinical diagnosis of USH1 in both eyes, meaning subjects with congenital profound deafness, vestibular dysfunction, and rod dystrophy, carrying biallelic class 4 or 5 variants in the MYO7A gene;
* Be affiliated with or beneficiary of a social security system (according to article L1121-8-1 of the French Public Health Code);

For participants in the MOST-VR mobility test and VR-ViSA visual search test (Streetlab), additional criteria apply:

* Sufficient knowledge of spoken and signed French to ensure understanding of tasks and instructions;
* Have a cochlear implant allowing comprehension of auditory instructions for the virtual reality mobility test and a MMSE score ≥ 20/25;
* Age between 18 and 75 years.

Exclusion Criteria:

* Unable to participate in all study visits;
* Expected to enter an experimental treatment trial at any time during this study;
* Presence of ocular conditions that may affect eye status other than retinitis pigmentosa (e.g., history of retinal detachment, glaucoma, vein occlusion, diabetic retinopathy, etc.);
* Participation in the previous gene replacement trial (USHSTAT, NCT01505062);
* Pregnant, delivering, or breastfeeding women (according to article L1121-5 of the French Public Health Code);
* Persons deprived of liberty by judicial or administrative decision (article L1121-6 of the French Public Health Code);
* Adults under legal protection measures or unable to provide consent (article L1121-8 of the French Public Health Code).

For participants in the MOST-VR mobility and VR-ViSA visual search tests, the following non-inclusion criteria apply:

* MMSE score without visual items ≤ 20/25;
* Physical or cognitive impairment that could interfere with mobility;
* Medication that may cause motor, visual, or cognitive disorders (e.g., APS, neuroleptics) or interfere with study assessments.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Usher syndrome (USB1B)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2032-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | The BCVA is assessed at Day 0 = initial visit, at Month 12, at Month 24, at Month 36 and Month 48 = end of the study. This assessment is taking 15 minutes.
  Change in visual acuity measured using the ETDRS scale over the course of the study.
Electroretinography (ERG) | The Retinal Degeneration Progression is assessed at Day 0 = initial visit, at Month 12, at Month 24, at Month 36 and Month 48 = end of the study. The ERG is taking 60 minutes.
  Evaluation of photoreceptor function decline assessed by electroretinography (ERG).
Full-field stimulus testing (FST) | The Retinal Degeneration Progression is assessed at Day 0 = initial visit, at Month 12, at Month 24, at Month 36 and Month 48 = end of the study. The FST is taking 90 minutes.
  Evaluation of photoreceptor function decline assessed by full-field stimulus testing (FST).

SECONDARY OUTCOMES:
Retinal Structure | The Retinal structure measurement is assessed at Day 0 = initial visit, at Month 12, at Month 24, at Month 36 and Month 48 = end of the study. The SD-OCT is taking 25 minutes.
  Changes in retinal morphology assessed by spectral-domain OCT (SD-OCT).
Fundus autofluorescence (FAF) | The Retinal structure measurement is assessed at Day 0 = initial visit, at Month 12, at Month 24, at Month 36 and Month 48 = end of the study. The FAF is taking 15 minutes.
  Changes in retinal morphology assessed by fundus autofluorescence (FAF).
OCT angiography (OCT-A) | The Retinal structure measurement is assessed at Day 0 = initial visit, at Month 12, at Month 24, at Month 36 and Month 48 = end of the study. The OCT-A is taking 25 minutes.
  Changes in retinal morphology assessed by OCT angiography (OCT-A).
Michigan Vision-Related Anxiety Questionnaire (MAVQ) | The Patient-reported outcomes is assessed at Day 0 = initial visit, at Month 12, at Month 24, at Month 36 and Month 48 = end of the study. The MAVQ is taking 30 minutes.
  Changes in vision-related anxiety and quality of life using the Michigan Vision-Related Anxiety Questionnaire (MAVQ).
Michigan Retinal Degeneration Questionnaire (MRDQ) | The Patient-reported outcomes is assessed at Day 0 = initial visit, at Month 12, at Month 24, at Month 36 and Month 48 = end of the study. The MRDQ is taking 30 minutes.
  Changes in vision-related anxiety and quality of life using the Michigan Retinal Degeneration Questionnaire (MRDQ).
MOST-VR (MObility Standardized Test in Virtual Reality) | The Functional Perfomance is assessed at Day 0 = initial visit, during Day 1 to Day 30 for reproductibility visits and at M24 (24 months). The MOST-VR is taking 75 minutes.
  Mobility search performance measured by Streetlab tests (MOST-VR).
VR-ViSA (Visual Search Assessment in Virtual Reality) | The Functional Perfomance is assessed at Day 0 = initial visit, during Day 1 to Day 30 for reproductibility visits and at Month 24. The VR-ViSA is taking 75 minutes.
  Visual search performance measured by Streetlab test (VR-ViSA).

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Audo, Pr, Principal Investigator — Centre National d'Ophtalmologie des Quinze-Vingts
Locations (1):
- Centre National d'Ophtalmologie des Quinze-Vingts, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT07278843/Prot_000.pdf